CLINICAL TRIAL: NCT03094949
Title: Comparison Between Laparoscopic Partial Nephrectomy and Ultrasound Guided Percutaneous Microwave Ablation for T1a Renal Tumor
Brief Title: Comparison Between Partial Nephrectomy and Ablation for Renal Tumor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Prof., Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 301jrcs
Record Dates: First submitted 2017-03-01; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Renal Cell Carcinoma
Keywords: microwave ablation; partial nephrectomy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partial Nephrectomy (Active Comparator): a kind of operation for renal tumor
  Interventions: Procedure: Partial Nephrectomy
- microwave ablation (Experimental): a kind of minimally invasive therapy by using microwave device for renal tumors
  Interventions: Procedure: microwave ablation

INTERVENTIONS:
Procedure: Partial Nephrectomy — The renal capsule is cut in a monopolar fashion around the tumor. After the renal artery is clamped with a bulldog clamp, cold cutting by scissors into the renal parenchymal boundary of the tumor is performed with an optimal surgical margin (a few millimeters). After retrograde injection of diluted indigo carmine, continuous suturing of the opened collecting system and transection of the major vessels is performed with intracorporeal knot-tying. Parenchymal suturing is performed in a continuous fashion. The 20-30 cm length of thread is used, and a knot is made at the end of the thread. A large Hem-o-lok polymer clip (Weck Closure System, Research Triangle Park, NC) is attached on the proximal side of the knot. Before the thread is tightened or cinched, the parenchyma is sutured in a running fashion with three or four stitches without any bolster so that the renal bed is kept in its natural position during the suturing.
  Arms: Partial Nephrectomy
Procedure: microwave ablation — Microwave ablation is a technique that uses thermal therapy to induce complete necrosis of tumor in situ by using microwave ablation device.Antenna in the microwave ablation device was percutaneously inserted into the tumor and placed at designated place under US guidance. For tumors less than 1.5 cm, one antenna was inserted and for tumors measuring 1.5 cm or greater, two antennae were inserted in parallel with an inter-antenna distance of 1.0-2.5 cm, which were used simultaneously during MWA to obtain larger ablation zone. A 20G thermocouple was inserted about 0.5-1 cm away from the tumor for real-time temperature monitoring during MWA. MW emission didn't stop until the heat-generated hyperechoic water vapor completely encompassed the entire tumor and the measured temperature reached 60°C or remained above 54°C for at least three minutes.
  Arms: microwave ablation

SUMMARY:
The therapeutic effectiveness of ultrasound guided cooled-probe microwave ablation and laparoscopic partial nephrectomy on T1a renal cell carcinoma is compared to find a better approach for renal tumor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the RCC of ≤4 cm maximum diameter were included in the study.

Exclusion Criteria:

* Patients having RCCs with vascular invasion, extrarenal spread or with benign renal tumors were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-07-01 (Actual); Primary Completion 2017-07-01 (Estimated); Study Completion 2017-09-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | 5 years
  using log-rank test

SECONDARY OUTCOMES:
local tumor progress(new lesion found adjacent to ablation zone) | 5 years
  using log-rank test
rate of intrarenal metastasis(new lesion found in the treated kidney, but not adjacent to ablation zone) | 5 years
  using log-rank test
rate of extrarenal metastasis(new lesion found outside of treated kidney) | 5 years
  using log-rank test
number of patients with side-effect and major complications | 1 month
  using chi-square test

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes